CLINICAL TRIAL: NCT01916889
Title: Validation Study of the 4-question "RACY"Delirium Screening Tool in General Medical In-patients From a Developing Country Setting
Brief Title: 4-question "RACY" Delirium Screening Tool Validation Study
Acronym: RACY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Jonathan Peter, Honorary Consultant, Department of Medicine, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCT 148/2013
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Delirium
Keywords: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RACY test (Experimental): 4-question "RACY" delirium screening tool
  Interventions: Other: RACY test

INTERVENTIONS:
Other: RACY test

SUMMARY:
Delirium is a serious medical condition associated with increased mortality, longer hospital stay, increased rates of institutionalisation, and declines in post-admission functionality. Despite the prognostic utility of diagnosing delirium and its utility as an important indicator of health quality in elderly patients in developed countries, it is not routinely screened for in many busy general medical in-patient settings, especially in developing countries. Unpublished data from a recent study of general medical in-patients in Groote Schuur Hospital, Cape Town, South Africa, found that no patients admitted during an 8-week period received any formal cognitive testing or had documentation of the presence/absence of delirium in routine clinical notes. This under-recognition is largely the result of the length and complexity of available delirium diagnostic tools e.g. Mini-mental state exam (MMSE), although the perceived lack of clinical importance and conflicting results about specific treatment modalities also contribute.

The investigators recently developed the simple 4-question "RACY" delirium screening tool for use in general medical in-patients. Preliminary data show the test to be simple and effective with a sensitivity and specificity of 78% and 85% respectively using a ROC-selected cut-point of RACY≤2. The investigators hypothesis that the RACY screening tool has the potential to be a simple and effective bedside delirium diagnostic instrument for use in non-geriatric, busy general medical in-patient settings. This study is a two-centre validation study to evaluate the diagnostic accuracy of this tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for admission to general medical wards (including within hospital transfer e.g. ICU discharge)
* >18 years and willing to give informed consent

Exclusion Criteria:

* Patient admitted directly to intensive care unit
* Patient refusing consent or <18 years old
* Patients unable to undergo delirium testing due to: i) Glasgow coma scale ≤ 12/15, ii) Aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1093 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (Sensitivity, specificity, likelihood ratios) of the "RACY" delirium screening tool | 48 hours
  The 4-question "RACY" delirium screening tool and reference delirium testing will be performed within 24 hours of hospital admission to the general medical wards. "RACY" delirium screening and reference delirium testing will be performed within 4 hours of each other by two independent testers. Testers performing the "RACY" delirium screening will be blinded to the results of the reference testing.

SECONDARY OUTCOMES:
12-month cognitive outcomes in patients <50 years | 12-months
  A subset of cohort patients <50 years diagnosed with delirium during acute general medical admission will undergo full neurocognitive assessment at 12-month post-enrolment.
Measurement of IL-6, IL-2, TNF-alpha, IFN-gamma, IGF-1, MCP-1, and hsCRP | 12-months
  Using samples stored at the time of delirium diagnosis, biomarker levels will be compared between delirium and non-delirium in-patients less than 50 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Peter, Principal Investigator — University of Cape Town; Peter Raubenheimer, Study Director — University of Cape Town
Locations (2):
- South Africa (2):
  - Groote Schuur Hospital, Cape Town
  - Victoria Hospital, Cape Town

REFERENCES:
- [Background] Stuart-Clark H, Vorajee N, Zuma S, Van Niekerk L, Burch V, Raubenheimer P, Peter JG. Twelve-month outcomes of patients admitted to the acute general medical service at Groote Schuur Hospital. S Afr Med J. 2012 May 23;102(6):549-53. doi: 10.7196/samj.5615. PMID 22668961